CLINICAL TRIAL: NCT06703619
Title: Comparative Evaluation of the Full Outline of UnResponsiveness (FOUR) Score and Glasgow Coma Scale in Predicting Clinical Outcomes in Patients With Altered Mental Status Presenting to the Emergency Department: A Prospective Cohort Study
Brief Title: Comparison Between GCS and FOUR Scores
Acronym: GCS/FOUR
Status: Completed | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20240520
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Coma
Keywords: GCS; FOUR score; COMA
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this observational study is to compare the predictive utility of the Full Outline of Unresponsiveness (FOUR) Score and the Glasgow Coma Scale (GCS) Score in determining outcomes among patients with altered mental status admitted to the emergency room. The main questions it aims to answer are:

Does the FOUR Score provide a more accurate prediction of patient outcomes than the GCS Score? Are there specific patient subgroups where one score is more effective than the other?

Participants will:

Undergo assessment of mental status using both the FOUR Score and the GCS Score during their emergency room admission.

Have their clinical outcomes monitored during their hospital stay.

DETAILED DESCRIPTION:
The Glasgow Coma Scale (GCS) is commonly used for neurological assessment, but it lacks the precision to cover the full range of consciousness changes.[1]

The GCS is a 15-point scale used to assess consciousness based on three components:

Eye Opening (E):

Spontaneous (4 points) To verbal command (3 points) To pain (2 points) No response (1 point)

Verbal Response (V):

Oriented (5 points) Confused (4 points) Inappropriate words (3 points) Incomprehensible sounds (2 points) No response (1 point)

Motor Response (M):

Obeys commands (6 points) Localizes pain (5 points) Withdrawal to pain (4 points) Abnormal flexion (decorticate posture, 3 points) Abnormal extension (decerebrate posture, 2 points) No response (1 point)

Scoring Range:

15 (best) to 3 (worst). A score ≤8 typically indicates severe brain injury. The Glasgow Coma Scale (GCS) cannot be applied to intubated or aphasic patients because their verbal responses cannot be assessed. Additionally, a withdrawal response to pain can easily be mistaken for a flexion response to pain. While eye-opening indicates wakefulness, it does not necessarily mean that the content of consciousness is intact, as seen in a persistent vegetative state. Furthermore, the GCS does not take into account important factors such as brainstem reflexes, changes in breathing patterns, or the need for mechanical ventilation, all of which could provide a clearer understanding of the coma's severity and offer a more comprehensive neurological assessment.[1-3]

Considering the limitations of the GCS, a new coma scale named the full outline of unresponsiveness (FOUR) score.[2] The scale has been designed to overcome the limitations mentioned above of GCS.

The FOUR score [2] completes it here as it has a higher neurological sophistication. The score is a 16-point scale consisting of four components: eye response, motor response, brainstem reflexes, and respiration.

Eye Response (E):

Eyelids open and tracking (4 points) Eyelids open but not tracking (3 points) Eyelids closed but open to loud voice (2 points) Eyelids closed and open only to pain (1 point) Eyelids closed with no response (0 points)

Motor Response (M):

Obeys commands (4 points) Localizes pain (3 points) Flexion to pain (2 points) Extension to pain (1 point) No response to pain (0 points)

Brainstem Reflexes (B):

Pupillary and corneal reflexes present (4 points) One reflex absent (3 points) Both reflexes absent (2 points) Pupillary reflex absent but corneal reflex present (1 point) No brainstem reflexes (0 points)

Respiration (R):

Not intubated, regular breathing (4 points) Not intubated, Cheyne-Stokes breathing (3 points) Not intubated, irregular breathing (2 points) Intubated and breathing above the ventilator rate (1 point) Intubated and apneic (0 points)

Scoring Range:

16 (best) to 0 (worst).

It can identify states of consciousness other than those approximated by GCS, such as vegetative state and locked-in state. It gives information in regard to respiratory drive and pattern and, therefore, can signal the necessity of mechanical ventilation in the comatose patient. It is more neurologically detailed by featuring brainstem reflexes and respiration components added to the test. It can also categorise the extent of the lowest value to three of the GCS. Hence, it is a more broad-based neurological exam that seems to have better potential to impact early definitive and triage.

Common clinical parameters used for evaluation and management in patients with altered mental status in the Iraqi setting are primarily focused on the use of the Glasgow Coma Scale (GCS) Score, which has been established to be of limited value in evaluating more complex neurological conditions. The Full Outline of Unresponsiveness (FOUR) Score has been proposed internationally as a more comprehensive tool, but its use and validation in the Iraqi population are relatively scarce. This absence of local studies on the comparison between the two scoring systems becomes a major concern as emergency patients may be at risk of the ways coaches devise strategies. The purpose of this study is to fill this gap by investigating and comparing the prognostic abilities of the FOUR Score and the GCS Score in Iraqi Emergency Room patients. Thus, the study aims at presenting information that may help decide when to implement better assessment tools that would ultimately improve patient care for those with the altered mental status.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency room with altered mental status.
* Patients were assessed using both the Full Outline of Unresponsiveness (FOUR) Score and the Glasgow Coma Scale (GCS) Score upon admission.
* Patients whose clinical outcomes (e.g., mortality, length of hospital stay, need for intensive care) are available for follow-up and analysis.

Exclusion Criteria:

* Patients with incomplete or missing data on FOUR and/or GCS assessments.
* Patients who leave against medical advice (LAMA) or are discharged before outcome data can be collected.
* Patients with pre-existing neurological conditions that might independently influence outcomes (e.g., severe dementia, long-standing neurodegenerative diseases).
* Patients in whom resuscitative measures were initiated but unsuccessful before scoring could be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients (aged 18 years and above) presenting to the emergency room with altered mental status due to various underlying conditions, such as traumatic brain injury, metabolic encephalopathy, stroke, or central nervous system infections.
  Participants will be selected from a tertiary care hospital emergency room where comprehensive medical and neurological assessments are routinely conducted. This population is expected to represent a diverse range of clinical presentations and severities of altered consciousness, making it suitable for evaluating the predictive performance of the Full Outline of Unresponsiveness (FOUR) score and the Glasgow Coma Scale (GCS).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
In hospital mortality | average of 10 days through discharge
  Mortality (death) during hospitalization
Accuracy Assessment of the Glasgow Coma Scale (GCS) | the first 12 hours after ER admission
  Glasgow Coma Scale (GCS): Range 3-15; higher scores indicate better neurological status.
Accuracy Assessment of the Full Outline of UnResponsiveness (FOUR) Score | the first 12 hours after ER admission
  Full Outline of Unresponsiveness (FOUR) score: Range 0-16; higher scores indicate better neurological status.

SECONDARY OUTCOMES:
Length of Hospitalization | average of 10 days through discharge
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Azeez Al-Hamadani, Professor of Neurology, Study Chair — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fischer M, Ruegg S, Czaplinski A, Strohmeier M, Lehmann A, Tschan F, Hunziker PR, Marsch SC. Inter-rater reliability of the Full Outline of UnResponsiveness score and the Glasgow Coma Scale in critically ill patients: a prospective observational study. Crit Care. 2010;14(2):R64. doi: 10.1186/cc8963. Epub 2010 Apr 14. PMID 20398274
- [Result] Wijdicks EF, Bamlet WR, Maramattom BV, Manno EM, McClelland RL. Validation of a new coma scale: The FOUR score. Ann Neurol. 2005 Oct;58(4):585-93. doi: 10.1002/ana.20611. PMID 16178024
- [Result] Segatore M, Way C. The Glasgow Coma Scale: time for change. Heart Lung. 1992 Nov-Dec;21(6):548-57. PMID 1447002